CLINICAL TRIAL: NCT05300373
Title: Prospective Observational Study Evaluating the Prevalence of Adenosine Deaminase (ADA) Enzyme Deficiency Disease in Patients With Lymphopenia and/or Immunoglobulin E Elevation in Adult Immunology and Hematology Clinics
Brief Title: Evaluation of Adenosine Deaminase (ADA) Enzyme Deficiency in Patients With Lymphopenia and/or Elevated Immunoglobulin E
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: TRPHARM (Industry)
Responsible Party: Sponsor
Other Study IDs: TR-ADA-009
Record Dates: First submitted 2022-03-18; First posted 2022-03-29 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Adenosine Deaminase Deficiency
Keywords: lymphopenia, adenosine deaminase, guithre paper
MeSH Terms: conditions — Severe combined immunodeficiency due to adenosine deaminase deficiency; Lymphopenia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: ADENOSINE DEAMINASE TEST — ADENOSINE DEAMINASE DEFICIENCY TEST

SUMMARY:
This study was designed as an observational, prospective, epidemiological screening study. Patients who have been admitted to the center and whose lymphopenia and/or Immunoglobulin E elevation has been detected in at least one examination in their medical history will be included.

In accordance with the relevant legislation, patients are required to accept and sign the Informed Consent Form regarding their participation in the study.

Current data that the physician has already questioned in his daily practice will be collected from patients who have agreed to participate in the study, and a blood sample will be taken from patients on Guthrie paper. This sample will be prepared by taking it from the patient as the physician deems appropriate, dripping it into a special area designated on Guthrie paper and drying it.

The test result will be sent to the researcher by e-mail. In case of formation of new information for each patient, consultation will be provided by the responsible researcher.

Thus, the prevalence of ADA enzyme deficiency disease in patients with lymphopenia will be evaluated. In addition, with this study, it will be scientifically demonstrated whether lymphopenia is a parameter that facilitates early diagnosis of ADA patients.

DETAILED DESCRIPTION:
Primary immunodeficiencies are encountered with signs and symptoms related to various disciplines of medicine and are detected more often in our country than in other societies.

Severe Combined Immunodeficiencies (SCID) are a heterogeneous group of diseases caused by hereditary errors in genes involved in the development and/or function of T, B, and sometimes NK cells, which cause serious dysfunction of the immune system. The incidence is estimated at 1/100,000 live births in the USA. Although the exact incidence of inbreeding is not known in our country, where inbreeding is common, it is expected that those who show autosomal recessive transition will be more common, especially. Each step that is effective in the emergence of an immune response creates the potential for a primary immunodeficiency disease. Due to the development of molecular and cellular techniques, the possibility of prenatal diagnosis has arisen with the detection of localization and mutations of the defective gene in various immunodeficiencies. The recognition of these disorders by clinicians is important for reducing long-term complications due to recurrent infections and preventing mortality with appropriate treatment.

The frequency of SCID in our country is unknown. Unlike in Europe and America, SCID types, which are autosomal recessive in our country, are considered to be the most common form due to the high rates of inbreeding. The figure obtained by comparing the number of live babies born in a year in Konya with the number of SCID cases diagnosed in the same year at the Pediatric Immunology Clinic of the Meram Faculty of Medicine of Selcuk University, the only primary immunodeficiency diagnostic center in the region, is 1/10,000. This preliminary study shows that in our country this disease is much more common than in Europe and America. About 1,300 a year in our country.considering that 000 babies have been born, it should be expected that 140 new cases of SCID should be encountered every year. The number of cases diagnosed in our country is much lower than this figure.

To date, more than 20 genetic defects have been identified that cause SCID. All known genetic defects disrupt the development of cells of the immune system, causing combined immunodeficiency. One of them, the ADA defect, is also a metabolic disease, due to which there is a lack of enzymes.

ADA catalyzes the deamination of purine nucleosides adenosine (Ado) and 2'-deoxyadenosine (dAdo), which are produced during the degradation and transformation of RNA and DNA. ADA is a cleansing enzyme; it detoxifies purines. In ADA deficiency, 2'-deoxyadenosine (dAdo) is phosphorylated and converted into deoxyadenosine triphosphate (dATP). Accumulation of DATP disrupts DNA repair and replication. In ADA deficiency, a high percentage of dATP accumulates, especially in erythrocytes and lymphocytes. Increased levels of adenosine break down the wall of the lymphocyte. It inhibits the development of lymphocytes in the thymus. A kind of lymphocyte intoxication occurs. It leads to a severe form of lymphopenia. Approximately 10-20% of AKIS are diagnosed as ADA enzyme deficiency. It shows an autosomal recessive transition. Your gene is 20. it is localized on the long arm of the chromosome.

Clinically, there are early and late onset types. Classic-early onset ADA deficiency: Although normal at birth, patients present with infections seen from the first months of life, resulting in death if left untreated. In addition to the SCI table, neuro-developmental disorders, sensorineural hearing loss and/or skeletal abnormalities have also been reported in these patients. Although hematopoietic stem cell transplantation, enzyme replacement therapy and gene therapy are treatment approaches that provide cure, early diagnosis determines the prognosis.

Late onset ADA deficiency: Patients may present with recurrent infections, autoimmunity, human papillomavirus (HPV) infections at an older age, even in adulthood. Lymphopenia is an invariable finding. High IgE and eosinophilia may be observed. In these cases, residual enzyme activity due to the type of mutation causes a late onset. This phenotype accounts for 10-15% of all cases of ADA deficiency.

Diagnosis: ADA enzyme deficiency is included in severe combined immunodeficiencies and is observed with lymphopenia and infections. The diagnosis is made by measuring the activity of the enzyme ADA in erythrocytes or lymphocytes in patients with suspected clinical and laboratory features (such as lymphopenia). By mutation analysis, a gene defect is shown. However, T-cell receptor excision circles (TREC) test is used for early diagnosis. However, since the TREC test is found to be normal at birth in late-onset patients, screening that leads patients to an early diagnosis can only be achieved by measuring ADA metabolites.

Although studies are continuing for SCID, which has not yet been included in the screening program in our country, the tandem mass spectrometer, which can be used to diagnose ADA deficiency, is used in newborn screening programs for metabolic diseases. Studies of newborn screening with a tandem mass spectrometer for ADA and PNP deficiencies, which is also a metabolic disease, began after 2010, and it has been shown that this method is a low-cost and reliable method. Early and late onset ADA deficiency cases can be detected with sensitivity and specificity reaching 100% with this method.

Importance of early diagnosis: In Early Onset ADA deficiency, patients usually consult a doctor with signs of infections. The fact that infections are already common in the dairy childhood age group makes diagnosis difficult. If there is no similar case in the family that has been diagnosed before, or if this is not paid attention to in the history, the diagnosis of the cases is delayed. In late-onset ADA deficiency, the diagnosis is much more difficult. Low awareness of the disease and its symptoms usually results in these cases not being diagnosed, not being able to get effective treatment, and organ damage. For this reason, early diagnosis is very important in terms of quality of life as well as vital importance.

ELIGIBILITY:
Inclusion Criteria:

1. Signing of the written informed consent form by the patient and/or his legal representative,

* The patient is between 18 and 40 years of age.
* Patients with one major and one minor criteria from the following criteria will be included in the study:

Major Criteria:

1. Lymphopenia: The patient has lymphopenia as a result of at least one hemogram,

   -The number of lymphocytes is below 1500/mm3
2. Immunoglobulin E height: The level of immunoglobulin E is above 120 kU/L.

Minor Criteria:

1. Two or more new ear infections within a year
2. Two or more new sinus infections within a year when there is no allergy
3. One pneumonia per year for more than a year
4. Chronic diarrhea with weight loss
5. Recurrent viral infections (Colds, herpes, warts, condyloma)
6. The need for repeated intravenous antibiotics to clear infections
7. Recurrent deep skin or internal organ abscesses
8. Persistent thrush or fungal infection of the skin or other place
9. Infection caused by tuberculosis-like bacteria that is normally harmless
10. Primary immunodeficiency in the family

Exclusion Criteria:

1. Having used drugs that can cause lymphopenia before being included in the study (chemotherapy, cytotoxic drug use, etc.),
2. The Ministry of Health COVID-19 diagnosis guide (nazofaringeal, nasal orofaringiyal or SARS-CoV-2 RNA PCR test and/or tomographic) as COVID-19, diagnosed and/or persons who had contact with patient recruitment criteria, patients diagnosed in this manner karsilasal PCR tests were negative even after those patients in the study will be taken.
3. Before being included in the study, it should be noted that other diseases that can cause lymphopenia (hematological diseases, oncological diseases, etc.) have been diagnosed with,
4. The patient has participated in an interventional clinical trial within the last 30 days,
5. Failure of the patient himself and/or his legal representative to give their consent to participate in the study,
6. According to the researcher's opinion, the patient will not be able to properly fulfill the study requirements,
7. Pregnancy and/or lactation period,
8. The fact that the volunteer participating in

Ages: 18 Years to 40 Years | Sex: All
Age Groups: Adult
Study Population: male and female patients aged 18-40 years
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-12-03 (Actual); Primary Completion 2022-01-03 (Actual); Study Completion 2023-12-03 (Estimated)

PRIMARY OUTCOMES:
The ratio of adult patients with immunoglobulin E elevation and/or lymphopenia who have an ADA metabolite test above the threshold value | 2 years
  The ratio of adult patients with immunoglobulin E elevation and/or lymphopenia who are above the ADA metabolite test threshold and are suspected of having ADA enzyme deficiency

SECONDARY OUTCOMES:
The relationship between of lymphopenia and ADA enzyme deficiency disease | 2 years
  The relationship between the level and frequency of lymphopenia and ADA enzyme deficiency disease
The relationship between lymphopenia and demographic parameters | 2 years
  The relationship between lymphopenia and demographic parameters
Family history and ADA | 2 years
  Family history of immunodeficiency/ADA
The existence of inbreeding | 2 years
  The existence of inbreeding
late ADA enzyme deficiency | 2 years
  The rate of late ADA enzyme deficiency disease
immunoglobulin E level and ADA enzyme deficiency | 2 years
  The relationship between immunoglobulin E level and ADA enzyme deficiency
infection frequency and ADA enzyme deciency | 2 years
  The relationship between infection frequency and ADA enzyme deficiency

CONTACTS AND LOCATIONS:
Locations (1):
- Konya Necmettin Erbakan University, Konya, Meram, Turkey (Türkiye)